CLINICAL TRIAL: NCT01493687
Title: A Phase 3 Randomized, Double Blind, 12 Week Vehicle Controlled, Parallel Group Study Assessing the Efficacy and Safety of CD5024 1 % Cream Versus Vehicle Cream in Subjects With Papulopustular Rosacea, Followed by a 40 Week Investigator Blinded Extension Comparing the Long Term Safety of CD5024 1% Cream Versus Azelaic Acid 15 % Gel.
Brief Title: Phase 3 Papulopustular Rosacea Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18170
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2015-01

CONDITIONS: Papulopustular Rosacea (PPR)
MeSH Terms: conditions — Rosacea | interventions — azelaic acid; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CD5024 (Experimental): CD5024 1% Cream
  Interventions: Drug: CD5024
- CD5024 Vehicle (Placebo Comparator): CD5024 Vehicle Cream
  Interventions: Drug: Azelaic acid 15% Gel

INTERVENTIONS:
Drug: CD5024 — CD5024 1% Cream, once daily
  Arms: CD5024
Drug: Azelaic acid 15% Gel — Topical Gel applied twice daily
  Arms: CD5024 Vehicle

SUMMARY:
The purpose of this study is to demonstrate that CD5024 1% cream is more effective than its vehicle when applied once daily, at bed time, during a 12 week period in subjects with Papulopustular Rosacea (PPR) and continues to be safe up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has papulopustular rosacea with an Investigator Global Assessment (IGA) score rated 3 (moderate) or 4 (severe),
2. The subject has at least 15 but not more than 70 inflammatory lesions (papules and pustules) on the face.

Exclusion Criteria:

1. The subject has particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other facial dermatoses that may be confounded with papulopustular rosacea, such as peri oral dermatitis, facial keratosis pilaris, seborrheic dermatitis, and acne,
2. The subject has rosacea with more than two nodules on the face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, M.D., Study Director — Galderma R&D, LLC
Locations (50):
- United States (40):
  - UAB Dermatology Clinical Research, Birmingham, Alabama
  - Northwest AR Clinical Trials Center, Rogers, Arkansas
  - Dermatology Research Associates, Los Angeles, California
  - University Clinical Trials, San Diego, California
  - Research Across America, Santa Ana, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - The Center for Clinical & Cosmetic Research, Aventura, Florida
  - The Dermatology and Aesthetic Center, Boca Raton, Florida
  - North Florida Dermatology Associates, Jacksonville, Florida
  - FXM Research Miramar, Miramar, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - The South Bend Clinic, LLP, South Bend, Indiana
  - Derm Research, PLLC, Louisville, Kentucky
  - Lawrence Green, MD, LLC, Rockville, Maryland
  - Henry Ford Health Systems Department of Dermatology, Detroit, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Central Dermatology PC, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Anderson & Collins Clinical Research,, Edison, New Jersey
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Department of Dermatology - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Dermatology Research Center of Cincinnati, Cincinnati, Ohio
  - Haber Dermatology Clinical Research Center, South Euclid, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Baker Allergy, Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - Palmetto Clinical Trial Services, LLC, Simpsonville, South Carolina
  - TriCities Skin and Cancer, Johnson City, Tennessee
  - Dermatology Associates of Kingsport, PC, Kingsport, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - PLLC dba Dermatology Associates, Seattle, Washington
  - The Polyclinic, Seattle, Washington
- Canada (10):
  - Stratica Medical Inc, Edmonton, Alberta
  - Derm Research@888 Inc., Vancouver, British Columbia
  - Dermadvances Research, Winnepeg, Manitoba
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Associates, Halifax, Nova Scotia
  - Skin Centre for Dermatology, Peterborough, Ontario
  - Toronto Research Centre, Inc., Toronto, Ontario
  - Windsor Clinical Research, Inc., Windsor, Ontario
  - Innovaderm Research. Inc, Montreal, Quebec
  - Siena Medical, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- CD5024 1% Cream: Part A & B: CD5024 1% Cream, once daily application
- CD5024 Vehicle Cream/Azelaic Acid 15% Gel: Part A: CD5024 Vehicle Cream, once daily application
  Part B: Azelaic acid 15% Gel, twice daily application
Period: Part A Vehicle Control (12 Weeks)
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream/Azelaic Acid 15% Gel
Started | 451 | 232
Completed | 414 | 210
Not Completed | 37 | 22
Not completed — Pregnancy | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 7 | 4
Not completed — Withdrawal by Subject | 18 | 7
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 7 | 8
Not completed — Other (noted on CRF) | 1 | 1
Period: Part B Long Term Active Control 40 Weeks
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream/Azelaic Acid 15% Gel
Started | 412 (414 completed Part A. Then 2 discontinued (lack of efficacy, subject request) prior to Part B.) | 210
Completed | 351 | 175
Not Completed | 61 | 35
Not completed — Pregnancy | 5 | 1
Not completed — Lack of Efficacy | 2 | 3
Not completed — Adverse Event | 5 | 4
Not completed — Withdrawal by Subject | 27 | 16
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 16 | 10
Not completed — Other (noted on eCRF) | 5 | 1
Period: Part C Safety Follow up (4 Weeks)
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream/Azelaic Acid 15% Gel
Started | 350 (351 completed Part B. Then 1 discontinued (subject request) prior to Part C.) | 175
Completed | 350 | 174
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- CD5024 1% Cream: Part A: CD5024 1% Cream, once daily application for 12 weeks Part B: CD5024 1% Cream, once daily application for 40 weeks
- CD5024 Vehicle Cream/Azelaic Acid 15% Gel: Part A: CD5024 Vehicle Cream, once daily application for 12 weeks
  Part B: Azelaic acid 15% Gel, twice daily application for 40 weeks
- Total: Total of all reporting groups
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream/Azelaic Acid 15% Gel | Total
Number analyzed (Participants) | 451 | 232 | 683
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (12.15) | 51.6 (11.92) | 50.4 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 152 | 466
  Male | 137 | 80 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 23 | 78
  Not Hispanic or Latino | 396 | 209 | 605
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 437 | 220 | 657
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Skin Photo Type [Number; unit: Participants] — DEFINITION OF SKIN PHOTOTYPE (T.B. Fitzpatrick):
  I: Always burns easily ; never tans II: Always burns easily ; tans minimally and with difficulty III: Burns minimally ; tans gradually and uniformly (light Brown) IV: Burns minimally ; always tans well (moderate brown) V: Rarely burns ; tans profusely (dark brown)) VI:Never burns ; deeply pigmented (black), tans profusely
  Participants
    I | 39 | 16 | 55
    II | 185 | 90 | 275
    III | 167 | 86 | 253
    IV | 51 | 26 | 77
    V | 8 | 11 | 19
    VI | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Percentage of subjects who achieve "Clear" (Score 0) or "Almost Clear" (Score 1) at Week 12 (ITT-LOCF) based on the Investigator Global Assessment (IGA) Score.
  Evaluation of papulopustular rosacea will be performed by the investigator based on the following 5 point scale:
  Clear = 0 (No inflammatory lesions present, no erythema); Almost Clear = 1 (Very few small papules/pustules, very mild erythema present); Mild = 2 (Few small papules/pustules, mild erythema); Moderate = 3 (Several small or large papules/pustules, moderate erythema); Severe = 4 (Numerous small and/or large papules/pustules, severe erythema)
Time Frame: Week 12
Population: LOCF, ITT
Measure: Number; unit: Percentage of participants
Groups:
- CD5024 1% Cream: CD5024: CD5024 1% Cream, once daily application for 12 weeks
- CD5024 Vehicle Cream: CD5024 Vehicle Cream, once daily application for 12 weeks
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream
Number analyzed (Participants) | 451 | 232
Percentage of participants | 38.4 | 11.6
Statistical Analysis 1: Comparison: CD5024 1% Cream vs CD5024 Vehicle Cream; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Absolute Change in Inflammatory Lesion Count
Description: Inflammatory lesion counts were conducted at each visit by the Investigator or study coordinator. Papules and pustules were counted separately on each of the five facial regions (forehead, chin, nose, right cheek, left cheek).
Time Frame: Baseline to Week 12
Population: LOCF, ITT
Measure: Mean (Standard Deviation); unit: Lesion count change
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream
Number analyzed (Participants) | 451 | 232
Lesion count change | -20.5 (15.95) | -12.0 (13.55)
Statistical Analysis 1: Comparison: CD5024 1% Cream vs CD5024 Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -8.13, 95% CI 2-sided [-10.12 to -6.13]

3. Secondary Outcome: Percent Change in Inflammatory Lesion Count From Baseline to Week 12 (ITT-LOCF)
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: LOCF, ITT
Measure: Mean (Standard Deviation); unit: Percentage of change in lesion counts
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream
Number analyzed (Participants) | 451 | 232
Percentage of change in lesion counts | -64.9 (39.91) | -41.6 (38.83)
Statistical Analysis 1: Comparison: CD5024 1% Cream vs CD5024 Vehicle Cream; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Time of signed informed consent to study end (~ 58 wks). Treatment emergent adverse events - occurred on date of 1st use of medication or after, except those reported from Day 1 lab data as blood sample was to be drawn before the time of 1st dose.
Groups:
- CD5024 1% Cream - Part A: Part A: CD5024 1% Cream, once daily application for 12 weeks
- CD5024 Vehicle Cream - Part A: Part A: CD5024 Vehicle Cream, once daily application for 12 weeks
- CD5024 1% Cream - Part B: Part B CD5024 1% Cream, once daily application for 40 weeks
- Azelaic Acid 15% Gel - Part B: Part B: Subjects in the CD5024 Vehicle Cream arm applied Azelaic Acid 15% Gel twice daily for 40 weeks
- CD5024 1% Cream - Part C; CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Part C: Part C: 4 week safety follow up. No drug applications
- CD5024 1% Cream - Overall; CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Overall: Overall number of subjects with adverse events for the entire duration of study
Arm/Group | CD5024 1% Cream - Part A | CD5024 Vehicle Cream - Part A | CD5024 1% Cream - Part B | Azelaic Acid 15% Gel - Part B | CD5024 1% Cream - Part C | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Part C | CD5024 1% Cream - Overall | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Overall
Serious Adverse Events (participants affected / at risk) | 3/452 | 1/231 | 7/412 | 8/210 | 0/350 | 1/175 | 10/452 | 9/232
Other Adverse Events (participants affected / at risk) | 30/452 | 10/231 | 93/412 | 47/210 | 4/350 | 0/175 | 110/452 | 52/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5024 1% Cream - Part A (N=452) | CD5024 Vehicle Cream - Part A (N=231) | CD5024 1% Cream - Part B (N=412) | Azelaic Acid 15% Gel - Part B (N=210) | CD5024 1% Cream - Part C (N=350) | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Part C (N=175) | CD5024 1% Cream - Overall (N=452) | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Overall (N=232)
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Oesophageal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhagic anaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD5024 1% Cream - Part A (N=452) | CD5024 Vehicle Cream - Part A (N=231) | CD5024 1% Cream - Part B (N=412) | Azelaic Acid 15% Gel - Part B (N=210) | CD5024 1% Cream - Part C (N=350) | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Part C (N=175) | CD5024 1% Cream - Overall (N=452) | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Overall (N=232)
Nasopharyngitis (Infections and infestations) | 12 | 6 | 54 | 31 | 1 | 0 | 63 | 34
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 31 | 14 | 2 | 0 | 37 | 16
Headache (Nervous system disorders) | 13 | 4 | 17 | 8 | 1 | 0 | 26 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submission for publication, presentation or use, the Institution and the Investigator shall submit in writing to the Contract Research Organization and Sponsor for review and comment any proposed oral or written publication, which period may be extended for an additional thirty (30) days if requested in writing by Contract Research Organization and Sponsor.